CLINICAL TRIAL: NCT00457613
Title: Effects of Alkaline Phosphatase on Renal Function in Patients With Severe Sepsis or Septic Shock.
Brief Title: Effects of Alkaline Phosphatase on Renal Function in Septic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP05
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2006-03

CONDITIONS: Severe; Septic; Shock
Keywords: alkaline phosphatase; sepsis; kidney function
MeSH Terms: conditions — Lymphoma, Follicular; Shock; Sepsis | interventions — Alkaline Phosphatase

INTERVENTIONS:
Drug: bolus injection, followed by a continuous infusion ( 24 h) (Alkaline phosphatase)

SUMMARY:
Septic shock is the most common cause of death in patients requiring intensive care. The kidney is one of the first organs to fail, stressing the importance to search for clinical interventions that may protect the kidneys during sepsis.

Alkaline phosphatase functions as a host defence molecule and is present in many cells and organs (e.g. intestine, placenta, liver, kidney and bone). Alkaline phosphatase has a dual mode of action. First, it binds to and, subsequently, dephosphorylates lipopolysaccharide (LPS). Second, the enzymatic reaction product monophosphoryl-LPS is a non-toxic substance for mammals which acts as a partial antagonist on the LPS receptor complex. In several animal studies, administration of alkaline phosphatase attenuates the inflammatory response and reduces mortality.

It is unknown whether these results can be extrapolated to septic patients . We studied the effects of alkaline phosphatse administration on kidney damage and function in patients with severe sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Proven or suspected Gram-negative bacterial infection
* Two out of four Systemic Inflammatory Response Syndrome (SIRS) criteria existing for less than 24 h
* Acute onset of end-organ dysfunction in the preceding 12 h

Exclusion Criteria:

* Prior therapy with alkaline phosphatase
* Known allergy for cow milk
* Probable death within 24 h
* Chronic renal failure requiring hemodialysis or peritoneal dialysis
* Acute pancreatitis with no established source of infection
* HIV seropositive
* Pregnant or lactating
* Confirmed Gram-positive or fungal sepsis
* Treatment with immunosuppressants including high doses of glucocorticosteroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-11; Study Completion 2006-03

PRIMARY OUTCOMES:
Biomarkers of kidney damage
kidney function
markers of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Study Director — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands